CLINICAL TRIAL: NCT03934424
Title: Exposure to Weight Stigmatization Content: Neural Correlations With Appetite Control, Social Support, Mood and Weight Stigma Experiences
Brief Title: Weight Stigma Effect on Neural Control of Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Katherene Anguah, Assistant Research Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013871
Record Dates: First submitted 2019-02-12; First posted 2019-05-01 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Appetitive Behavior
Keywords: appetite; fMRI; overweight; obese; weight stigma
MeSH Terms: conditions — Appetitive Behavior; Overweight; Obesity; Weight Prejudice

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to read a weight stigma article or control article and subsequently scanned for fMRI data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Stigma (Experimental): Weight stigma, read a weight stigma article for 5-10 minutes on one day
  Interventions: Behavioral: Weight stigma
- Ethnic stigma (Other): Ethnic stigma, read an ethnic stigma article for 5-10 minutes on one day
  Interventions: Behavioral: Ethnic stigma

INTERVENTIONS:
Behavioral: Weight stigma — Subject will read an article depicting discrimination against individuals with higher body weights for 5-10 minutes on one day
  Arms: Weight Stigma
Behavioral: Ethnic stigma — Subject will read a control article for weight stigma depicting discrimination against individuals from a minority ethnic group for 5-10 minutes on one day
  Arms: Ethnic stigma

SUMMARY:
The limited data available suggest that exposure to weight-based stigmatization leads to overeating and increased desire for food. In the present study, overweight and obese individuals (BMI from 25-35 kg/m2) who are generally healthy will be randomized to read a weight-stigma article or control article and subsequently scanned to collect fMRI data. These procedures will be employed to accomplish two specific aims.

Specific Aim 1: Determine the neural mechanisms involved in exposure to weight stigma on central control of appetite in overweight and obese individuals. To accomplish this aim we will collect fMRI data in study participants when viewing food and scenery pictures after being exposed to either a weight-stigma or control article. In addition, participants will complete validated questionnaires to measure perceived weight-stigma experiences and social support for eating and physical activity. Hypothesis: After reading an article depicting weight stigmatization, when shown pictures of food in the fMRI scanner, overweight/obese individuals that perceive themselves as having experienced higher levels of weight stigma and lower levels of social support, will have higher activations of brain regions that control appetite and food reward (amygdala, orbitofrontal cortex, striatum, insula) and reduced activations in brain areas that regulate self-control and decision making (prefrontal cortex and cingulate cortex respectively) compared to a control group that reads a non-weight stigma article.

Specific Aim 2: To assess the relationship between activity in appetitive and self-control brain regions and self-reported, eating-related behavior. To accomplish this aim, participants will also complete questionnaires that measure self-reported food intake motivation (dietary restraint, disinhibition and hunger), appetitive responses, and mood. Hypothesis: Higher activations in appetite and reward regions and lower activations in self-control brain regions will be correlated with higher levels of dietary disinhibition, hunger/appetite, and dietary restraint.

DETAILED DESCRIPTION:
Introduction Over two-thirds of Americans are either overweight or obese (Fryar et al., 2016) and thus the search for therapeutic strategies for the overweight/obesity epidemic is key. As much as 20% of overweight/obese individuals also report having weight stigma experiences (Levy and Pilfer, 2012) and may experience stigmatization repeatedly over the course of their lifetimes. Weight stigma, as defined by Araiza and Wellman (Araiza and Wellman, 2017), is the social depreciation and condemnation of individuals with higher body weight.

Emerging data from two recent review articles demonstrate that the negative impact of weight stigma experienced by overweight and obese individuals occurs on the physiological, psychological, and behavioral levels (Vartanian and Porter, 2016; Wu and Berry, 2018). Weight stigma could actually lead to overconsumption of food and eating disorders such as binge eating (Wott and Carels, 2010; Almeida et al., 2011) which can further exacerbate the obesity epidemic. For example, the more participants perceived themselves as experiencing weight stigma, the more calories they selected (Araiza and Wellman, 2017) or consumed (Major et al., 2014) and the more poorly they performed on cognitive tests (Araiza and Wellman, 2017) when they read an article depicting discrimination against individuals with higher body weight compared to a control group. In the Major et al. study, women who perceived themselves as being overweight consumed 80 calories more of a high-calorie snack which translated to a magnitude of effect of 47%. Perceived weight stigma has also been shown to be positively correlated with emotional and rigid restrained eating as well as predicting weight gain over a ten-week period (Wellman et al., 2017).

Importantly, individuals with higher body weights are more affected when put in situations that remind them more of weight stigmatization (Major et al., 2014; Hunger et al., 2015), though not everyone may respond in the same manner. While data exist to show the negative impacts of weight stigma of overweight/obese individuals on eating behavior, there is a paucity of data regarding the effect of exposure to weight-stigma content on the neural control of appetite and self-control in overweight/obese individuals. The so-called 'appetitive network' is centered around the following interconnected brain regions: the amygdala and hippocampus, the orbitofrontal cortex (OFC) and adjacent ventromedial prefrontal cortex (VMPFC), the striatum, and the insula. These areas of the brain are normally activated during functional magnetic resonance imaging (fMRI) studies where food cue reactivity is assessed, and the activity is regulated by peripheral signals of energy balance, current hunger, and personality traits (Dagher, 2012). Furthermore, how these neural control measures correlate with self-reports of weight stigma experiences, social support for eating behavior and physical activity, food intake motivation (dietary restraint, disinhibition and hunger), mood and appetite require further investigation.

Study Design This is a cross-sectional study of overweight/obese, generally healthy subjects. After having completed a telephone prescreening test to determine eligibility for the study, subjects will be invited to the Brain Imaging Center (BIC) at the University of Missouri for a one-time research visit lasting approximately three hours. The subject will report to the BIC in the fasted state. The sequence of events during this test visit is outlined in Figure 1 and is described in detail below.

Upon arrival at the BIC, the subject will be screened for eligibility for MRI research following the standard University of Missouri screening protocol. The subject will then be taken through the informed consent process and then testing will begin. Informed consent is performed in a quiet, closed office and the subject will be given ample time to discuss the study and ask questions. Anthropometric measurements (weight and height), as well as a finger prick glucose measurement, is preformed and subsequently, the subject is asked to fill out a series of questionnaires (appetite/ mood, social support, weight stigma experiences, Three-Factor Eating questionnaire). Research staff are present to answer any questions the subject may have about the surveys. Then, the subject will read their assigned weight-stigma or control article (randomization to either the control or weight stigma article condition will be done before data collection commence). One of the questionnaires (appetite/mood) is repeated after reading the article just prior to scanning, and also again after scanning is over. The subject then undergoes fMRI scanning followed by a final repeat of the appetite/mood survey and a finger stick for glucose measurement. Upon completion of all the test procedures, the subject is debriefed as to the purpose of the article and told that the article was fictional.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals aged from 18 to 55 years
* BMI 25-35 kg/m2 will be recruited

Exclusion Criteria:

* Being on a weight-loss or special diet
* Taking any medications or drugs known to affect appetite
* Have serious claustrophobia.
* Individuals with mental disorders (self-report) will be excluded.
* Due to MRI, any individuals with metallic objects in their body, including surgical staples left in the body following surgery, middle ear prosthesis, permanent eye liner, metal foreign objects lodged inside the eye, heart pacemakers, and/or pins inside the knee or other joints or who are pregnant or could be pregnant (assessed through a urine pregnancy test for women) will be excluded from this study because of the risk associated with the MRI scanner.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow in appetite/reward regions | ~1 hour
  BOLD contrast-Measures activity in the brain by detecting changes in cerebral blood flow
Change in cerebral blood flow on self-control regions | ~ 1 hour
  BOLD contrast-Measures activity in the brain by detecting changes in cerebral blood flow
Score of perceived appetite | Time 0, before and after fMRI scanning
  Scale of 1 to 100 with higher scores indicating greater appetite

SECONDARY OUTCOMES:
Score of Dietary Restraint | Baseline
  Scale of 0-21, with higher score indicating higher restraint
Score of Disinhibition | Baseline
  Scale of 0 to 16, with higher score indicating greater disinhibition
Score of perceived Hunger | Baseline
  Scale of 0 to 14, with higher score indication higher hunger level
Score of Weight stigma experience | Baseline
  scale of 1 to 7 with higher scores indicating greater stigma experiences
Score of Social support | Baseline
  Scale of 1 to 5 for each question
Glucose | Time 0 and at the end of fMRI scanning
  mg/dL
Frequency of weight stigma experience | Baseline
  scale of 0 to 9 with higher scores indicating greater frequency of stigma experiences

CONTACTS AND LOCATIONS:
Overall Officials: Katherene O Anguah, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy BR, Pilver CE. Residual stigma: psychological distress among the formerly overweight. Soc Sci Med. 2012 Jul;75(2):297-9. doi: 10.1016/j.socscimed.2012.03.007. Epub 2012 Apr 3. PMID 22560867
- [Background] Araiza AM, Wellman JD. Weight stigma predicts inhibitory control and food selection in response to the salience of weight discrimination. Appetite. 2017 Jul 1;114:382-390. doi: 10.1016/j.appet.2017.04.009. Epub 2017 Apr 14. PMID 28416329
- [Background] Vartanian LR, Porter AM. Weight stigma and eating behavior: A review of the literature. Appetite. 2016 Jul 1;102:3-14. doi: 10.1016/j.appet.2016.01.034. Epub 2016 Jan 29. PMID 26829371
- [Background] Wu YK, Berry DC. Impact of weight stigma on physiological and psychological health outcomes for overweight and obese adults: A systematic review. J Adv Nurs. 2018 May;74(5):1030-1042. doi: 10.1111/jan.13511. Epub 2017 Dec 8. PMID 29171076
- [Background] Wott CB, Carels RA. Overt weight stigma, psychological distress and weight loss treatment outcomes. J Health Psychol. 2010 May;15(4):608-14. doi: 10.1177/1359105309355339. PMID 20460417
- [Background] Almeida L, Savoy S, Boxer P. The role of weight stigmatization in cumulative risk for binge eating. J Clin Psychol. 2011 Mar;67(3):278-92. doi: 10.1002/jclp.20749. Epub 2010 Dec 3. PMID 21254056
- [Background] Blodorn A, Major B, Hunger J, Miller C. Unpacking the psychological weight of weight stigma: A rejection-expectation pathway. J Exp Soc Psychol. 2016 Mar 1;63:69-76. doi: 10.1016/j.jesp.2015.12.003. PMID 26752792
- [Background] Wellman JD, Araiza AM, Newell EE, McCoy SK. Weight stigma facilitates unhealthy eating and weight gain via fear of fat. Stigma Health. 2018 Aug;3(3):186-194. doi: 10.1037/sah0000088. Epub 2017 Feb 9. PMID 30221195
- [Background] Hunger JM, Major B, Blodorn A, Miller CT. Weighed down by stigma: How weight-based social identity threat contributes to weight gain and poor health. Soc Personal Psychol Compass. 2015 Jun;9(6):255-268. doi: 10.1111/spc3.12172. Epub 2015 Jun 4. PMID 29225670
- [Background] Dagher A. Functional brain imaging of appetite. Trends Endocrinol Metab. 2012 May;23(5):250-60. doi: 10.1016/j.tem.2012.02.009. Epub 2012 Apr 5. PMID 22483361
- See also: Prevalence of overweight, obesity, and extreme obesity among adults aged 20 and over — https://www.cdc.gov/nchs/data/hestat/obesity_adult_13_14/obesity_adult_13_14.htm